CLINICAL TRIAL: NCT06046326
Title: Evaluate the Effectiveness of a Virtual Community of Practice Via a Web-based Application Versus Individual and Self-administered Online Education to Improve the Activation of Middle-aged People with Multimorbidity.
Brief Title: Evaluate the Effectiveness of a Virtual Community of Practice
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI22/01124
Record Dates: First submitted 2023-06-22; First posted 2023-09-21 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Chronic Diseases
Keywords: Chronic Diseases; Virtual community of practice empowerment
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- virtual community of practice (Experimental): The intervention group will be offered participation for 12 months in a VCoP based ona gamified web-based application.
  Interventions: Behavioral: virtual community of practice
- control group (No Intervention): The control group will receive individual, content-focused education through a web platform that will cover the same topics as the VCoP but will be self-administered and without social interaction within theplatform.

INTERVENTIONS:
Behavioral: virtual community of practice — The intervention group will be offered participation for 12 months in a VCoP based ona gamified web-based application.
  Arms: virtual community of practice

SUMMARY:
Objective: To evaluate and compare the effectiveness and cost-effectiveness of a Virtual Community of Practice (VCoP) via a web-based application versus individual and self-administered online education to improve the activation of middle-aged people with multimorbidity.

Design: Randomized controlled pragmatic clinical trial with two parallel arms and 18 months follow-up.

Setting: Primary health centres and hospitals (Catalonia, Madrid, and the Canary Islands). Population: Middleaged people (30-60 years old) with multimorbidity (≥=2 chronic diseases). Sample size: 240 patients.

Randomization: all participants will be randomly assigned to the intervention (VCoP) or the active control group. Data analysis will be blinded to intervention allocation. Intervention: The intervention group will be offered participation for 12 months in a VCoP based on a gamified web-based application. The control group will receive individual, content-focused education through a web platform that will cover the same topics as the VCoP but will be self-administered and without social interaction within the platform.

Measurements: The main variable will be measured using the Patient Activation Measure (PAM) questionnaire at baseline, 6, 12 and 18 months. Secondary variables: participant sociodemographics, depression (PHQ-9), anxiety (HADS-A), treatment burden (TBQ), quality of life (EQ-5D-5L), variables related to the use of health resources and to the use of the VCoP. Analysis: Mixed-effects linear regression will be used to determine the effects of the VCoP on the changes in patient activation. Scores at baseline, 6, 12 and 18 months will be included as a fixed effect variable, and the patient and health professional as random effect variables. Analyses will be performed on an intention-to-treat basis. An economic evaluation will be carried out to analyze the cost-effectiveness of the VCoP compared to active control, from the National Health System and social perspectives.

DETAILED DESCRIPTION:
Objective: To evaluate and compare the effectiveness and cost-effectiveness of a Virtual Community of Practice (VCoP) via a web-based application versus individual and self-administered online education to improve the activation of middle-aged people with multimorbidity.

Design: Randomized controlled pragmatic clinical trial with two parallel arms and 18 months follow-up.

Setting: Primary health centres and hospitals (Catalonia, Madrid, and the Canary Islands). Population:

Inclusion criteria:

* Age between 30 and 60 years
* diagnosis of ≥ 2 chronic diseases
* have a computer with an Internet connection or another mobile device (tablet or smartphone)
* be able to follow the requirements of the study have signed the informed consent

Exclusion criteria:

* Low probability of cooperation in the study
* with a terminal illness, physical or mental disability that prevents answering the questionnaires correctly
* Sample size: 240 patients.

Randomization: all participants will be randomly assigned to the intervention (VCoP) or the active control group. Data analysis will be blinded to intervention allocation.

Intervention: The intervention group will be offered participation for 12 months in a VCoP based on a web-based application. The control group will receive individual, content-focused education through a web platform that will cover the same topics as the VCoP but will be self-administered and without social interaction within the platform.

Measurements:

participant sociodemographics variables The main variable will be measured using the Patient Activation Measure (PAM) questionnaire at baseline, 6, 12 and 18 months. It consists of 13 items that assess people´s Knowledge, skills and confidence in self-care for their health and medical care, measured using a 1-4 likert scale with a total score that is transferred to a scale between 0 and 100.

Secondary variables:

Patient Health Questionnaire at baseline, 6, 12 and 18 months It is a short instrument, designed to be self-administered. It consists of 9 items that evaluate the presence of depressive symptoms present in the last 2 weeks. Each item has a severity index: 0 = "never", 1 = "some days", 2 = "more than half of the days" and 3 = "almost every day". The puntuation is between 0 and 27 (worse puntuation).

Hospital Anxiety and Depression Scale at baseline, 6, 12 and 18 months It is a 14-item questionnaire composed of two sub-scales (HAD-A: anxiety and HAD-D: depression), of 7 items each that are scored from 0 to 3. The puntuation is between 0 and 21 (worse puntuation). The authors recommend points of 8 for possible cases and >10 for probable cases on both subscales.

Treatment Burden Questionnaire at baseline, 6, 12 and 18 months It is a questionnaire of 13 items that uses a Likert scale that ranges from 0 (not a problem) to 20 (it is an important problem) and that assesses the burden related to taking medication, self-care, laboratory tests, medical appointments, the need for organization, administrative tasks, compliance with diet and physical activity and the social impact of treatment. The puntuation is between 0 and 260 (worse puntuation).

European quality of life. Euroqol-5D at baseline, 6, 12 and 18 months Assesses health-related quality of life (HRQoL) both in the general population and in groups of patients with different pathologies. It comprises 5 dimensions (mobility, self-care, activities of daily living, pain/discomfort, and anxiety/depression). Each dimension has 3 items that are scored from 1, no problems, to 3, many problems. There is a visual analogue scale that scores from 0 (worst health status imaginable) to 100 (best health status imaginable)

Analysis: Mixed-effects linear regression will be used to determine the effects of the VCoP on the changes in patient activation. Scores at baseline, 6, 12 and 18 months will be included as a fixed effect variable, and the patient and health professional as random effect variables.

Analyses will be performed on an intention-to-treat basis. An economic evaluation will be carried out to analyze the cost-effectiveness of the VCoP compared to active control, from the National Health System and social perspectives.

ELIGIBILITY:
Inclusion Criteria:

* Middleagedpeople (30-60 years old)
* with multimorbidity (≥=2 chronic diseases).

Exclusion Criteria:

* Low probability of cooperation in the study
* situation of transients or displaced persons, institutionalized, with some terminal illness, physical or mental disability that prevents them from answering the questionnaires correctly.
* When the contact telephone number/email is not available in the CAP/hospital database.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 30 - 60 years old
Enrollment: 240 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
the Patient Activation Measure (PAM) | Baseline
  It consists of 13 items that assess people's knowledge, skills, and confidence in self-care for their health and medical care, measured using a 1-4 Likert scale with a total score that is transferred to a scale between 0 and 100.
the Patient Activation Measure (PAM) | 12 months
  It consists of 13 items that assess people's knowledge, skills, and confidence in self-care for their health and medical care, measured using a 1-4 Likert scale with a total score that is transferred to a scale between 0 and 100.
the Patient Activation Measure (PAM) | 18 months
  It consists of 13 items that assess people's knowledge, skills, and confidence in self-care for their health and medical care, measured using a 1-4 Likert scale with a total score that is transferred to a scale between 0 and 100.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 | Baseline
  It is a short instrument, designed to be self-administered. It consists of 9 items that evaluate the presence of depressive symptoms present in the last 2 weeks. Each item has a severity index: 0 = "never", 1 = "some days", 2 = "more than half of the days" and 3 = "almost every day". The puntuation is between 0 and 27 (worse puntuation).
Patient Health Questionnaire-9 | 12 months
  It is a short instrument, designed to be self-administered. It consists of 9 items that evaluate the presence of depressive symptoms present in the last 2 weeks. Each item has a severity index: 0 = "never", 1 = "some days", 2 = "more than half of the days" and 3 = "almost every day". The puntuation is between 0 and 27 (worse puntuation).
Patient Health Questionnaire-9 | 18 months
  It is a short instrument, designed to be self-administered. It consists of 9 items that evaluate the presence of depressive symptoms present in the last 2 weeks. Each item has a severity index: 0 = "never", 1 = "some days", 2 = "more than half of the days" and 3 = "almost every day". The puntuation is between 0 and 27 (worse puntuation).
Hospital Anxiety and Depression Scale (HADS) | Baseline
  It is a 14-item questionnaire composed of two sub-scales (HAD-A: anxiety and HAD-D: depression), of 7 items each that are scored from 0 to 3. The puntuation is between 0 and 21 (worse puntuation). The authors recommend points of 8 for possible cases and >10 for probable cases on both subscales.
Hospital Anxiety and Depression Scale (HADS) | 12 months
  It is a 14-item questionnaire composed of two sub-scales (HAD-A: anxiety and HAD-D: depression), of 7 items each that are scored from 0 to 3. The puntuation is between 0 and 21 (worse puntuation). The authors recommend points of 8 for possible cases and >10 for probable cases on both subscales.
Hospital Anxiety and Depression Scale (HADS) | 18 months
  It is a 14-item questionnaire composed of two sub-scales (HAD-A: anxiety and HAD-D: depression), of 7 items each that are scored from 0 to 3. The puntuation is between 0 and 21 (worse puntuation). The authors recommend points of 8 for possible cases and >10 for probable cases on both subscales.
Treatment Burden Questionnaire-TBQ | Baseline
  It is a questionnaire of 13 items that uses a Likert scale that ranges from 0 (not a problem) to 20 (it is an important problem) and that assesses the burden related to taking medication, self-care, laboratory tests, medical appointments, the need for organization, administrative tasks, compliance with diet and physical activity and the social impact of treatment. The puntuation is between 0 and 260 (worse puntuation). on the self-administered Treatment Burden Questionnaire - TBQ
Treatment Burden Questionnaire-TBQ | 12 months
  It is a questionnaire of 13 items that uses a Likert scale that ranges from 0 (not a problem) to 20 (it is an important problem) and that assesses the burden related to taking medication, self-care, laboratory tests, medical appointments, the need for organization, administrative tasks, compliance with diet and physical activity and the social impact of treatment. The puntuation is between 0 and 260 (worse puntuation). on the self-administered Treatment Burden Questionnaire - TBQ
Treatment Burden Questionnaire-TBQ | 18 months
  It is a questionnaire of 13 items that uses a Likert scale that ranges from 0 (not a problem) to 20 (it is an important problem) and that assesses the burden related to taking medication, self-care, laboratory tests, medical appointments, the need for organization, administrative tasks, compliance with diet and physical activity and the social impact of treatment. The puntuation is between 0 and 260 (worse puntuation). on the self-administered Treatment Burden Questionnaire - TBQ
European quality of life-5 dimensions. E5-5D-5L questionnaire | Baseline
  Assesses health-related quality of life (HRQoL) both in the general population and in groups of patients with different pathologies. It comprises 5 dimensions (mobility, self-care, activities of daily living, pain/discomfort, and anxiety/depression). Each dimension has 3 items that are scored from 1, no problems, to 3, many problems. There is a visual analogue scale that scores from 0 (worst health status imaginable) to 100 (best health status imaginable)
European quality of life-5 dimensions. E5-5D-5L questionnaire | 12 months
  Assesses health-related quality of life (HRQoL) both in the general population and in groups of patients with different pathologies. It comprises 5 dimensions (mobility, self-care, activities of daily living, pain/discomfort, and anxiety/depression). Each dimension has 3 items that are scored from 1, no problems, to 3, many problems. There is a visual analogue scale that scores from 0 (worst health status imaginable) to 100 (best health status imaginable)
European quality of life-5 dimensions. E5-5D-5L questionnaire | 18 months
  Assesses health-related quality of life (HRQoL) both in the general population and in groups of patients with different pathologies. It comprises 5 dimensions (mobility, self-care, activities of daily living, pain/discomfort, and anxiety/depression). Each dimension has 3 items that are scored from 1, no problems, to 3, many problems. There is a visual analogue scale that scores from 0 (worst health status imaginable) to 100 (best health status imaginable)

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Gerencia Asistencial Atención Primaria, Madrid, Madrid
  - González Atención González, Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Campillejo A, Gefaell-Larrondo I, Ramos-Garcia V, Koatz D, Santos-Alvarez A, Barrio-Cortes J, Gomez-Rueda S, Calderon-Larranaga A, Cifuentes P, Company-Sancho C, Dominguez-Coello S, Garcia-Garcia FJ, Garrido-Elustondo S, Gonzalez de Leon B, Ramon-Vazquez J, Martin C, Suarez-Fernandez C, Parra-Caballero P, Vicente-Rabaneda EF, Quiroga-Colina P, Ramirez-Puerta AB, Ruiz-Lopez M, Tello-Bernabe ME, Sanchez-Gamborino E, Ugalde-Abiega B, Vall-Roque H, Duarte-Diaz A, Abt-Sacks A, Hernandez-Yumar A, Torres-Castano A, Alvarez-Perez Y, Muth C, van den Akker M, Montori VM, Orrego C, Perestelo-Perez L, Gonzalez-Gonzalez AI. Implementation of a virtual community of practice to promote the empowerment of middle-aged people with multimorbidity: study protocol of a randomised controlled trial. BMJ Open. 2024 May 24;14(5):e084937. doi: 10.1136/bmjopen-2024-084937. PMID 38803252